CLINICAL TRIAL: NCT04313907
Title: Use of Low Intensity Laser Combined With Topical Clonazepam for the Treatment of Burning Mouth Syndrome
Brief Title: Low Level Laser Therapy Plus Topical Clonazepam Treatment to Burning Mouth Symdrome
Acronym: BurnLasCLo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Elba Rosa Leyva Huerta, Professor full time, PhD, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIE/0505/02/2019
Record Dates: First submitted 2020-03-06; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Burning Mouth Syndrome
Keywords: low-level laser therapy; topical clonazepam
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Low-Level Light Therapy; Clonazepam

STUDY DESIGN:
Intervention Model Description: group 1:active laser+topical clonazepam, group 2:inactive laser+topical clonazepam, group 3:active laser+placebo clonazepam
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acitve laser+topical clonazepam (Experimental): Using active laser (six sesions) 980 nm, 14 j , plus topical clonazepam 1 mg, 3 times at day, same 14 days both
  Interventions: Combination Product: low level laser therapy plus topical clonazepam
- Sham laser+topical clonazepam (Sham Comparator): Using sham laser (six sesions) plus topical clonazepam 1 mg, 3 times at day, same 14 days both
  Interventions: Drug: Sham laser plus topical clonazepam
- Active laser+placebo of topical clonazepam (Placebo Comparator): Using active laser (six sesions) 980 nm, 14 j , plus placebo of topical clonazepam (lactose), 3 times at day, same 14 days both
  Interventions: Radiation: Active laser plus placebo of topical clonazepam

INTERVENTIONS:
Combination Product: low level laser therapy plus topical clonazepam — combination of treatment, low level laser therapy (15 joules, 6 sesions, 14 days) plus topical clonazepam (1 mg,3 times per day, 14 days)
  Arms: Acitve laser+topical clonazepam
Drug: Sham laser plus topical clonazepam — Sham laser therapy (0 joules, 6 sesions, 14 days) plus topical clonazepam(1 mg,3 times per day, 14 days)
  Arms: Sham laser+topical clonazepam
Radiation: Active laser plus placebo of topical clonazepam — low level laser therapy (15 joules, 6 sesions, 14 days) plus placebo topical clonazepam(lactose,3 times per day, 14 days)
  Arms: Active laser+placebo of topical clonazepam

SUMMARY:
Burning mouth syndrome (BMS) is a condition that affects the oral mucosa; this is seen mainly in postmenopausal women. The intensity of burning and its clinical manifestations may be variable between patients. The etiology of the BMS is unknown, just as it is the therapeutic; hence the latter has not been fully accepted. Therefore, the use of low-level laser therapy (LLLT) and topical clonazepam have been proposed as treatment alternatives. The objective is to assess the effectiveness of the combination of LLLT and topical clonazepam for the reduction of burning symptoms. Three groups will be randomly formed: 1) the first group will received topical clonazepam therapy (half of a 2 mg tablet), patients in this group will be asked to applied it in a mouthwash type for 3 minutes and then spit it out; to the same group, six sessions of LLLT (Biolase 10 ©) will be applied in every second day intervals; 2) the second group, will received the same treatment with clonazepam and laser therapies with similar characteristics to the study group, but the laser will be deactivated; 3) the third group, will receive six sessions of LLLT (Biolase 10 ©) in every second day intervals and placebo tablets with similar characteristics to those of clonazepam. For all groups, both treatments will be received for two weeks. For the assessment of oral burning the visual analog scale (VAS) and the Oral Health Impact Profile-14 (OHIP-14) will be used; with these tools we will measure how oral disorders affect daily life. The measurement scales will be applied at the initial assessment and at day 14th, one month, two months and three months post treatment. The means obtained to assess the effectiveness of the treatment will be compared.

DETAILED DESCRIPTION:
The study will be carried out at the oral medicine clinic of the Division of Postgraduate Studies and Research of the Faculty of Dentistry of the National Autonomous University of Mexico, during the period of August 2019 to June 2020. This research was approved by the Ethics and Research Committee of the Faculty of Dentistry - Universidad Nacional Autonoma de Mexico. Inclusion criteria will be all patients with BMS, indistinctively of gender. The sample size will be 10 patients in each group, calculated using PaaS computer program with a power of 90.552% to reject the null hypothesis; based on the literature where an average difference of 4 points was obtained in the visual analogue scale from 8.0 to 4.0 with a standard deviation of 1.5 for the group that used laser and 3.0 for the control group, with a significance level of 0.05, in this calculation a number of 9 participants were obtained and the final group size was calculated adding a loss of 10%.

Initially, the patient will be assessed by an oral medicine resident and professor. If abnormalities of the mucosa are observed during the assessment, the patient will undergo blood and microbiological tests or biopsy according to the suspected diagnosis; if a diagnosis of BMS is confirmed, the patient will be invited to be part of the study.

Using a computer program, randomized block allocation was performed to guarantee equitable participation in each group. Closed envelopes will be used, each envelope will contain the information of which group each patient belongs to and the measurement tools (questionnaires EVA and OHIP-14) that will be applied at the initial moment, at 14 days, 1 month, 2 months and 3 months post treatment.

On an individual basis, all patients included in the study will be explained how to use and apply topical clonazepam or placebo tablets, which the patient must suck for 3 minutes periods, after their meals, trying to pass it through all the oral areas; the treatment must not be swallowed nor be placed exclusively under the tongue; to later spit out the leftovers. The tablets corresponding to the days between each laser application will be delivered and the application maneuvers of topical clonazepam or placebo will be evaluated on the morning of the application of the laser treatment, the corresponding observations will be made if necessary. A form with the instructions will be delivered.

Patients will be applied Biolase brand InGaAsp diode laser, wavelength 940 nm, tip 400 um, with applications in 10 sites in the oral cavity [lateral of tongue (2 sites), jugal mucosa, lower lip and floor of the mouth) bilaterally at a distance of 15 mm, 10 seconds per point, 15 joules each poit. If the patient reports other specific places where he perceives burning symptoms, it will be applied at the site and the information will be collected for inclusion in the results. Sham laser group will be applying laser inactive therapy with the same specifications. They will carry out 6 sessions, for the same 2 weeks that the topical treatment will last.

This research is in according with the regulations of the general health law regarding health research and is at greater than minimum risk.

ELIGIBILITY:
Inclusion Criteria:

* Burning mouth sensation without oral lesions that could be involved with painful symptoms
* Symtoms of burning sensation more than 3 months

Exclusion Criteria:

* Patients who are under antineoplastic treatment or with a history of malignant neoplasms of the head and neck
* Active treatment with benzodiazepines or systemic antidepressants
* Pregnant women
* Patients unable to follow the indications for administration of oral topical medications
* Unstimulated saliva production ≤ 0,1 mililiters/minute
* Sistemic diseases that can produce burning sensation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-06-16 (Estimated); Study Completion 2020-10-16 (Estimated)

PRIMARY OUTCOMES:
Burning Sensation | Change from baseline of Burning sensation using Visual Analogue Scale at 15 days, 1 month, 2 months, 3 months.
  Visual Analogue Scale using scale from 0 (No burning sensation) to 10 (maximum burning sensation)

SECONDARY OUTCOMES:
Quality of life- Oral Health Impact Profile | Change from baseline of Quality of life using OHIP-14 at 15 days, 1 month, 2 months, 3 months.
  Oral Health Impact Profile short form of 14 questions, 7 dimensions. Values from 0 to 56, value of 0 is better quality of life and 56 very poor quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Division de Estudios de Posgrado e Investigacion en Odontologia, Universidad Nacional Autonoma de Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] dos Santos Lde F, de Andrade SC, Nogueira GE, Leao JC, de Freitas PM. Phototherapy on the Treatment of Burning Mouth Syndrome: A Prospective Analysis of 20 Cases. Photochem Photobiol. 2015 Sep-Oct;91(5):1231-6. doi: 10.1111/php.12490. Epub 2015 Aug 4. PMID 26138316
- [Result] Minor JS, Epstein JB. Burning mouth syndrome and secondary oral burning. Otolaryngol Clin North Am. 2011 Feb;44(1):205-19, vii. doi: 10.1016/j.otc.2010.09.008. PMID 21093630
- [Result] Kisely S, Forbes M, Sawyer E, Black E, Lalloo R. A systematic review of randomized trials for the treatment of burning mouth syndrome. J Psychosom Res. 2016 Jul;86:39-46. doi: 10.1016/j.jpsychores.2016.05.001. Epub 2016 May 9. PMID 27302545
- [Result] Heckmann SM, Kirchner E, Grushka M, Wichmann MG, Hummel T. A double-blind study on clonazepam in patients with burning mouth syndrome. Laryngoscope. 2012 Apr;122(4):813-6. doi: 10.1002/lary.22490. Epub 2012 Feb 16. PMID 22344742
- [Result] Romeo U, Del Vecchio A, Capocci M, Maggiore C, Ripari M. The low level laser therapy in the management of neurological burning mouth syndrome. A pilot study. Ann Stomatol (Roma). 2010 Jan;1(1):14-8. Epub 2010 Jun 29. PMID 22238700
- [Result] Valenzuela S, Lopez-Jornet P. Effects of low-level laser therapy on burning mouth syndrome. J Oral Rehabil. 2017 Feb;44(2):125-132. doi: 10.1111/joor.12463. Epub 2016 Dec 22. PMID 27893167
- [Result] Al-Maweri SA, Javed F, Kalakonda B, AlAizari NA, Al-Soneidar W, Al-Akwa A. Efficacy of low level laser therapy in the treatment of burning mouth syndrome: A systematic review. Photodiagnosis Photodyn Ther. 2017 Mar;17:188-193. doi: 10.1016/j.pdpdt.2016.11.017. Epub 2016 Dec 2. PMID 27919663
- [Result] Gremeau-Richard C, Woda A, Navez ML, Attal N, Bouhassira D, Gagnieu MC, Laluque JF, Picard P, Pionchon P, Tubert S. Topical clonazepam in stomatodynia: a randomised placebo-controlled study. Pain. 2004 Mar;108(1-2):51-7. doi: 10.1016/j.pain.2003.12.002. PMID 15109507
- [Result] Arbabi-Kalati F, Bakhshani NM, Rasti M. Evaluation of the efficacy of low-level laser in improving the symptoms of burning mouth syndrome. J Clin Exp Dent. 2015 Oct 1;7(4):e524-7. doi: 10.4317/jced.52298. eCollection 2015 Oct. PMID 26535101
- [Result] Arduino PG, Cafaro A, Garrone M, Gambino A, Cabras M, Romagnoli E, Broccoletti R. A randomized pilot study to assess the safety and the value of low-level laser therapy versus clonazepam in patients with burning mouth syndrome. Lasers Med Sci. 2016 May;31(4):811-6. doi: 10.1007/s10103-016-1897-8. Epub 2016 Feb 12. PMID 26873501
- [Result] Sugaya NN, Silva EF, Kato IT, Prates R, Gallo CB, Pellegrini VD. Low Intensity laser therapy in patients with burning mouth syndrome: a randomized, placebo-controlled study. Braz Oral Res. 2016 Oct 10;30(1):e108. doi: 10.1590/1807-3107BOR-2016.vol30.0108. PMID 27737361
- [Result] Spanemberg JC, Lopez Lopez J, de Figueiredo MA, Cherubini K, Salum FG. Efficacy of low-level laser therapy for the treatment of burning mouth syndrome: a randomized, controlled trial. J Biomed Opt. 2015 Sep;20(9):098001. doi: 10.1117/1.JBO.20.9.098001. PMID 26359814